CLINICAL TRIAL: NCT01746472
Title: Online Social Networks for Dissemination of Smoking Cessation Interventions
Brief Title: Study of the Diffusion of a Smoking Cessation Application Through an Online Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 1R01CA155369-01A1 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2015-03

CONDITIONS: Use and Dissemination of Smoking Cessation Intervention; Cessation of Smoking
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- 2 - B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition B-passive
- 3 - B-active (Experimental)
  Interventions: Behavioral: Facebook app - condition B-active
- 4 - B-active, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition B-active; Behavioral: Facebook app - condition B-passive
- 6 - z, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition z; Behavioral: Facebook app - condition B-passive
- 7 - z, B-active (Experimental)
  Interventions: Behavioral: Facebook app - condition z; Behavioral: Facebook app - condition B-active
- 8 - z, B-active, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition z; Behavioral: Facebook app - condition B-active; Behavioral: Facebook app - condition B-passive
- 10 - t, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition B-passive
- 11 - t, B-active (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition B-active
- 12 - t, B-active, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition B-active; Behavioral: Facebook app - condition B-passive
- 14 - t, z (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition z
- 15 - t, z, B-active (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition z; Behavioral: Facebook app - condition B-active
- 16 - t, z, B-active, B-passive (Experimental)
  Interventions: Behavioral: Facebook app - condition t; Behavioral: Facebook app - condition z; Behavioral: Facebook app - condition B-active; Behavioral: Facebook app - condition B-passive

INTERVENTIONS:
Behavioral: Facebook app - condition t — Application components hypothesized to increase the duration (t, time) that a participant spends using the application.
  Arms: 10 - t, B-passive; 11 - t, B-active; 12 - t, B-active, B-passive; 14 - t, z; 15 - t, z, B-active; 16 - t, z, B-active, B-passive
Behavioral: Facebook app - condition z — Application components hypothesized to increase the number of friends that a user has that are eligible to install the application.
  Arms: 14 - t, z; 15 - t, z, B-active; 16 - t, z, B-active, B-passive; 6 - z, B-passive; 7 - z, B-active; 8 - z, B-active, B-passive
Behavioral: Facebook app - condition B-active — Application components hypothesized to increase the contagiousness of the app by increasing a users ability and desire to proactively contact others.
  Other Names: Ba
  Arms: 11 - t, B-active; 12 - t, B-active, B-passive; 15 - t, z, B-active; 16 - t, z, B-active, B-passive; 3 - B-active; 4 - B-active, B-passive; 7 - z, B-active; 8 - z, B-active, B-passive
Behavioral: Facebook app - condition B-passive — Application components hypothesized to increase the contagiousness of the app by increasing the passive diffusion of information from the user to their friends.
  Other Names: Bp
  Arms: 10 - t, B-passive; 12 - t, B-active, B-passive; 16 - t, z, B-active, B-passive; 2 - B-passive; 4 - B-active, B-passive; 6 - z, B-passive; 8 - z, B-active, B-passive

SUMMARY:
Effective evidence-based interventions exist for smoking cessation delivered over the Internet, but consumer acceptance and adherence remains low. Scalable and efficient mechanisms to disseminate these interventions online are needed, and existing online social networks provide a potential mechanism. This is a proposal for a randomized, factorial trial of the dissemination of an evidence-based intervention through the massive Facebook social network, with the goal of determining intervention characteristics that drive viral spread.

ELIGIBILITY:
Inclusion Criteria:

* Facebook user
* Age 18 years or older
* Entered UbiQUITous Facebook Application
* Confirms smoker status
* U.S. resident

Exclusion Criteria:

* Non-smoker
* Under 18 years old
* Non-U.S. resident
* Non-Facebook advertisement point of entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11413 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reproductive rate | 30 days
  The investigators will measure the reproductive rate for each condition, in other words the average number of additional individuals that install the application for each original individual recruited to participate. Higher reproductive rates indicate more efficient and faster dissemination.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Graham, PhD, Principal Investigator — Truth Initiative
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Cobb NK, Jacobs MA, Saul J, Wileyto EP, Graham AL. Diffusion of an evidence-based smoking cessation intervention through Facebook: a randomised controlled trial study protocol. BMJ Open. 2014 Jan 21;4(1):e004089. doi: 10.1136/bmjopen-2013-004089. PMID 24448847
- See also: UbiQUITous Facebook Application (Intervention) — http://apps.facebook.com/quitlab/?utm_source=clinicaltrials.gov